CLINICAL TRIAL: NCT02334436
Title: A Phase III, Multi-center, Randomized, Double Blind, Placebo-controlled, Single Dose, Trial to Demonstrate the Safety and Efficacy of DWP-450 in Adult Subjects for Treatment of Moderate-to-severe Glabellar Lines
Brief Title: A Phase III Study to Demonstrate the Safety and Efficacy of DWP-450 to Treat Glabellar Lines - EV-002
Acronym: EV-002
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Evolus, Inc. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EV-002
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — Botulinum Toxins, Type A; DWP450; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum toxin, Type A (Experimental): Botulinum toxin, Type A
  Interventions: Biological: Botulinum toxin, Type A
- Placebo (Placebo Comparator): 0.9% sterile, unpreserved saline
  Interventions: Other: 0.9% sterile, unpreserved saline

INTERVENTIONS:
Biological: Botulinum toxin, Type A — Botulinum toxin, Type A
  Other Names: DWP-450 (Botulinum purified neurotoxin, Type A) Injection; DWP-450
  Arms: Botulinum toxin, Type A
Other: 0.9% sterile, unpreserved saline — Placebo Comparator Arm
  Arms: Placebo

SUMMARY:
The primary objective is to demonstrate the safety and efficacy of DWP-450 (Botulinum purified neurotoxin, Type A) Injection in the treatment of moderate to severe glabellar lines associated with corrugator and/or procerus muscle activity in adult subjects

DETAILED DESCRIPTION:
Three hundred and twenty-four eligible subjects will be randomly assigned 3:1 to receive DWP-450 or placebo. Safety and efficacy will be assessed on Days 2, 7, 14, 30, 90, 120 and 150. The primary efficacy end point assesses the effectiveness of the DWP-450 against placebo on Day 30 in a superiority design.

ELIGIBILITY:
Inclusion Criteria:

* Subjects is an adult, of at least 18 years of age
* Subject is able to provide informed consent and comply with study instructions
* Subject has moderate to severe glabellar lines at maximum frown as assessed by the investigator using the GLS
* Subject has moderate to severe glabellar lines at maximum frown as assessed by the subject using the GLS
* Subject is willing and able to complete the entire course of the study

Exclusion Criteria:

* Previous treatment with botulinum toxin of any serotype in any area within the last 6 months
* Previous treatment with any facial aesthetic procedure (e.g. injection with fillers, chemical peeling, photo rejuvenation) in the glabellar area within the last 12 months
* Previous insertion of permanent material in the glabellar area
* Planned treatment with botulinum toxin of any serotype in any other body region during the study period
* Any surgery in the glabellar area including surgical removal of the corrugator, procerus, or depressor supercilii muscles or a combination of these, or scars in the glabellar area and the surrounding areas (including eye brow)
* Energy-based or cryo-therapy based treatment of facial muscles superior to the lateral canthus
* Any other planned facial aesthetic procedure during the trial period, superior to the level of the lateral canthus (subjects can continue with their usual skin care routine)
* Subjects who may not respond to 20 Units of botulinum toxin (e.g., inability to substantially lessen glabellar frown lines even by physically spreading them apart)
* Marked facial asymmetry
* Ptosis of eyelid and/or eyebrow, or history of eyelid and/or eyebrow ptosis
* History of facial nerve palsy
* Excessive dermatochalasis, deep dermal scarring, thick sebaceous skin
* Any active infection in the area of the injection sites
* Medical condition that may affect neuromuscular function (e.g., myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis)
* Evidence of recent alcohol or drug abuse
* Medical or psychiatric conditions that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study
* Pregnant or sexually active female subjects who are of childbearing potential and who are not willing to use an acceptable form of contraception
* Known allergy or hypersensitivity to botulinum toxin preparation
* Participation in another interventional clinical study within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rui Avelar, MD, Study Director — Evolus, iInc.
Locations (1):
- The Clinical Testing Center of Beverly Hills, Beverly Hills, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin, Type A | Placebo
Started | 246 | 78
Completed | 237 | 77
Not Completed | 9 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin, Type A | Placebo | Total
Number analyzed (Participants) | 246 | 78 | 324
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 219 | 72 | 291
  >=65 years | 27 | 6 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (11.54) | 50.4 (10.14) | 51.2 (11.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 220 | 70 | 290
  Male | 26 | 8 | 34

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a ≥2 Point Improvement in Glabellar Line Scale (GLS) as Independently Assessed by Investigator and and Subject
Description: The primary efficacy end point assesses the effectiveness of DWP-450 against placebo on Day 30. The primary efficacy measure is a composite end point. Using the GLS scale, investigators and subjects will assess the glabellar lines at Day 0 and Day 30. A subject is a responder only if both the investigator and subject independently agree that a ≥2 improvement has occurred from Day 0 to Day 30.
  GLS is scored: 0=none, 1=mild, 2=moderate, 3=severe.
Time Frame: Day 30
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Botulinum Toxin, Type A | Placebo
Number analyzed (Participants) | 240 | 75
percentage of responders | 70.4 [64.2 to 76.1] | 1.3 [0.0 to 7.2]

2. Secondary Outcome: Percentage of Participants With a ≥2 Point Improvement in Glabellar Line Scale (GLS) as Independently Assessed by Investigator and and Subject
Description: Secondary endpoint was the proportion of subjects classified as responders on Day 90. This was a composite endpoint based on both the Investigator and subject assessments of glabellar lines at maximum frown on the GLS; a subject was a responder only if both the Investigator and subject independently agreed that a ≥2 point improvement had occurred from Day 0 to 90 Day.
  GLS is scored: 0=none, 1=mild, 2=moderate, 3=severe.
Time Frame: 90 Days
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Botulinum Toxin, Type A | Placebo
Number analyzed (Participants) | 233 | 76
percentage of responders | 25.8 [20.3 to 31.9] | 0.0 [0.0 to 4.7]

3. Secondary Outcome: Percentage of Participants With a ≥2 Point Improvement in Glabellar Line Scale (GLS) as Independently Assessed by Investigator and and Subject
Description: Secondary endpoint was the proportion of subjects classified as responders on Day 120. This was a composite endpoint based on both the Investigator and subject assessments of glabellar lines at maximum frown on the GLS; a subject was a responder only if both the Investigator and subject independently agreed that a ≥2 point improvement had occurred from Day 0 to 120 Day
  GLS is scored: 0=none, 1=mild, 2=moderate, 3=severe.
Time Frame: Day 120
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Botulinum Toxin, Type A | Placebo
Number analyzed (Participants) | 233 | 75
percentage of responders | 12.4 [8.5 to 17.4] | 0.0 [0.0 to 4.8]

4. Secondary Outcome: Percentage of Participants With a ≥2 Point Improvement in Glabellar Line Scale (GLS) as Independently Assessed by Investigator and and Subject
Description: Secondary endpoint was the proportion of subjects classified as responders on Day 150. This was a composite endpoint based on both the Investigator and subject assessments of glabellar lines at maximum frown on the GLS; a subject was a responder only if both the Investigator and subject independently agreed that a ≥2 point improvement had occurred from Day 0 to 150 Day
  GLS is scored: 0=none, 1=mild, 2=moderate, 3=severe.
Time Frame: Day 150
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Botulinum Toxin, Type A | Placebo
Number analyzed (Participants) | 237 | 77
percentage of responders | 4.6 [2.3 to 8.2] | 0.0 [0.0 to 4.7]

ADVERSE EVENTS:
Arm/Group | Botulinum Toxin, Type A | Placebo
Serious Adverse Events (participants affected / at risk) | 4/246 | 0/78
Other Adverse Events (participants affected / at risk) | 66/246 | 21/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botulinum Toxin, Type A (N=246) | Placebo (N=78)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stress-induced cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botulinum Toxin, Type A (N=246) | Placebo (N=78)
Headache (Nervous system disorders) | 21 (28) | 7 (7)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1)
Eyelid edema (Eye disorders) | 2 (2) | 0 (0)
Mild wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 4 (4) | 0 (0)
Mild dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0)
Dysesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 1 (1) | 0 (0)
Restless leg syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (4) | 0 (0)
Asthenopia (Eye disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Eyebrow ptosis (Eye disorders) | 2 (2) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 3 (3) | 0 (0)
Injection site pain (General disorders) | 2 (2) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Adnexa uteri mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menstrual disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Glucose urine present (Investigations) | 1 (1) | 0 (0)
Diabetes mellitis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Spinal decompression (Surgical and medical procedures) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth abcess (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin sensitization (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No